CLINICAL TRIAL: NCT02233972
Title: A Drug-Drug Interaction Study To Investigate The Ginkgolides Meglumine Injection To Alter The Pharmacokinetics Of Midazolam.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Z-YXPU-ZS-IV5
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-08

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics; Ginkgolides Meglumine Injection
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam and Ginkgolides Meglumine Injection (Experimental): Midazolam: tablet, 7.5 mg. Midazolam will be taken on Day 1 and Day 22. Ginkgolides Meglumine Injection: 25mg, intravenous drip, once a day. It will be used on Day 8 -Day 21, 14 days totally.
  Interventions: Drug: Midazolam; Drug: Ginkgolides Meglumine Injection
- Midazolam and placebo (Placebo Comparator): Midazolam: tablet, 7.5 mg. Midazolam will be taken on Day 1 and Day 22. Placebo: Sodium Chloride Injection, 250 ml, intravenous drip, once a day. It will be used on Day 8 -Day 21, 14 days totally.
  Interventions: Drug: Midazolam; Drug: placebo

INTERVENTIONS:
Drug: Midazolam
Drug: Ginkgolides Meglumine Injection
  Arms: Midazolam and Ginkgolides Meglumine Injection
Drug: placebo
  Arms: Midazolam and placebo

SUMMARY:
This is an open label, randomized, Parallel Assignment, placebo-controlled study. One of the purposes of this study is to investigate the multiple dosing Ginkgolides Meglumine Injection to alter the pharmacokinetics of Midazolam, the other is to calculate the pharmacokinetic parameters after Single and multiple dosing of Ginkgolides Meglumine Injection.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-40.
* Male.
* Subjects have standard weight( generally not less than 50 kg), and body mass index (BMI) within 19-25.
* All physical examinations( including ECG, kidney function, liver function, blood routine, urine routines, etc) are normal.
* Subjects have no history of significant diseases, allergy or orthostatic hypotension.
* All subjects sign the informed consent after being informed all possible adverse drug reaction and .are able to complete all examination defined.

Exclusion Criteria:

* Subjects who cannot communicate with medical staff, and subjects with cerebral insufficiency or psychological problem.
* Partner of subjects have plan to pregnant.
* Subject have primary disease in vital organ.
* Subjects have a history of drug dependence or psychosis in last 2 years.
* Subjects with severe blood loss or blood donation more than 200 mL in the prior 3 months.
* Subjects who have participated in another clinical trial within the prior 3 months.
* Known or suspected to have a history of alcohol or drug abuse.
* Subjects who have abnormal clinical significance after checking preclinical laboratory data and physical examinations.
* Known allergy to pharmaceutical ingredient of Ginkgolides Meglumine Injection or allergy sufferers who are allergic to more than two kinds of food or drugs in the past.
* Subjects who have used any drugs in the prior 2 weeks.
* Subjects have unexplained infections.
* The subjects could not complete the study in the opinion of the Principal Investigator due to any reason.
* Subjects who test positive at screening for human immunodeficiency virus (HIV), hepatitis C virus (HCV) , hepatitis B surface antigen (HbsAg), etc.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters：Cmax、Tmax、AUC0-24h、T1/2、CL/F、Vz/F for Midazolam. | Day 1 and Day 22
Pharmacokinetics parameters：AUC0-24h（Day 22/ Day 1）、Cmax（Day 22/ Day 1）for Midazolam. | Day 1 and Day 22
Pharmacokinetics parameters：Cmax、Tmax、AUC0-24h、T1/2、CL/F、Vz/F for Ginkgolides Meglumine Injection. | Day 8
Pharmacokinetics parameters：T1/2、CL/F、Vz/F、Cmax,ss、Cmin,ss、Cav,ss、Tmax,ss、AUCtau,ss for Ginkgolides Meglumine Injection. | Day 19 and Day22
Pharmacokinetics parameters: Racc for Ginkgolides Meglumine Injection. | Day 19

SECONDARY OUTCOMES:
Safety assessments will be based on adverse event reports and the results of vital sign measurements, electrocardiogram, electrocardiograph monitoring and clinical laboratory tests. | Day 0, Day 1, Day 8-22 and Day 23
  Adverse event reports will be assessed at Day1, Day 8-22, Day 23. Vital sign measurements will be assessed at Screening stage, Day 0, Day 1, Day 8-22, Day 23. Electrocardiogram monitoring will be assessed at Day 1, Day 8-22. Clinical laboratory tests will be assessed at Screening stage and Day 23. Electrocardiogram will be assessed at Screening stage, Day 0, Day 8-22 and Day 23

CONTACTS AND LOCATIONS:
Overall Officials: Ou Ning, Principal Investigator — First Affiliated Hospital of Nanjing Medical University (Jiangsu Province Hospital)
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjing, Jiangsu, China